CLINICAL TRIAL: NCT06100003
Title: A Real-world Observational Clinical Study Aims to Assess the Consistency of Clinical Efficacy in Gastric Cancer Treatment and Drug Susceptibility Outcomes Using a Novel Drug Susceptibility Testing Method
Brief Title: A Clinical Study Aims to Assess the Consistency of Clinical Efficacy in Gastric Cancer Treatment and Drug Susceptibility Outcomes Using a Novel Drug Susceptibility Testing Method
Status: Recruiting | Type: Observational
Sponsor: Funan Liu (Other)
Collaborators: Institute of Health and Medical Technology, Hefei Institutes of Physical Science, Chinese Academy of Sciences (Unknown); Precedo Pharmaceuticals Co. Ltd. (Unknown); Suzhou Institute of Biomedical Engineering and Technology, Chinese Academy of Sciences, Suzhou 215163, China (Unknown)
Responsible Party: Sponsor-Investigator, Funan Liu, professor, China Medical University, China
Organization: China Medical University, China (Other)
Other Study IDs: ZKPRS-CMU1H-01
Record Dates: First submitted 2023-10-07; First posted 2023-10-25 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Gastric Cancer; Organoids
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a real-world observational clinical study. Patients diagnosed as gastric cancer through histopathology were screened and enrolled. Before anti-tumor treatment, gastroscopy biopsy tissue specimens, surgical specimens, and malignant pleural effusion or ascites specimens, etc. are collected. The investigators will perform a drug sensitivity testing based on a novel drug susceptibility testing method to test the commonly used anti-tumor treatment regimens. Patients were given conventional anti-tumor treatment according to the medical judgment of the doctors. Finally, the investigator will evaluate the consistency of clinical efficacy in gastric cancer treatment and drug susceptibility outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 and ≤80;
2. Patients with gastric cancer diagnosed by histopathology;
3. Patients who need neoadjuvant treatment; adjuvant therapy after radical surgery or palliative treatment;
4. Fresh tumor tissue specimens or malignant pleural effusion or ascites can be obtained;
5. Patients who sign the informed consent form, and are able to comply with the study period treatment process.

Exclusion Criteria:

1. Inability to follow the research protocol;
2. Inability to obtain relevant fresh specimens by biopsy/surgery/puncture;
3. Concomitant contraindications to chemotherapy;
4. pregnant or lactating women;
5. Patients deemed inappropriate by investigators.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with gastric cancer in the First Affiliated Hospital of China Medical University
Sampling Method: Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | From date of surgery until the date of first documented recurrence，up to 3 years
  An Indicator of efficacy of postoperative adjuvant therapy
Sensitivity | Through study completion, an average of 1 year
  Cases in which drug susceptibility results are sensitive to the antineoplastic regimen as a percentage of the cases that are effective in clinical evaluation
Specificity | Through study completion, an average of 1 year
  Cases in which drug susceptibility results are resistance to the antineoplastic regimen as a percentage of the cases that are ineffective in clinical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Zhenning Wang, doctor, Principal Investigator — The First Affiliated Hospital of China Medical Univeristy; Funan Liu, doctor, Principal Investigator — The First Affiliated Hospital of China Medical Univeristy
Locations (1):
- Phase I Clinical Trials Center Of The First Hospital of China Medical University, Shenyang, Liaoning, China